CLINICAL TRIAL: NCT06964139
Title: Learning Curve Associated With Hydrus Microstent Implantation
Brief Title: Hydrus Learning Curve Study
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Craig Chaya, Assistant Professor (Clinical), University of Utah
Other Study IDs: 180462
Record Dates: First submitted 2025-03-21; First posted 2025-05-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Surgery; Surgical Procedures, Minimally Invasive; Training; Training Effectiveness; Learning Curve

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Fellows: Glaucoma surgical fellows with minimal surgical experience
  Interventions: Other: Surgical video grading

INTERVENTIONS:
Other: Surgical video grading — Videos of fellow surgical cases will be randomized in sequence and provided to a masked grader who will review cases and record primary and secondary endpoints.

SUMMARY:
The goal of this observational study is to better understand the learning curve among novice glaucoma surgeons performing Hydrus microstent insertion. The main question it aims to answer is what is the average number of cases does it take new glaucoma surgical fellows to become competent in Hydrus insertion. Researchers will review and grade videos of surgical cases. Participating fellows will complete a survey reporting the number of cases they had completed before beginning their glaucoma surgical fellowship and how many Hydrus cases they performed during their fellowship before they felt comfortable performing Hydrus cases without an attending surgeon overseeing their work.

ELIGIBILITY:
Inclusion Criteria:

* Current glaucoma fellow at the Moran Eye Center, Washington University or Baylor University

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Glaucoma fellow at the Moran Eye Center, Washington University or Baylor University
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Mean number of cases across all fellows needed to achieve and maintain at least an 80% competence score | through study completion, an average of 9 months
  The competency matrix for Hydrus follows recommended surgical procedural steps. There are 12 competency steps that will be scored on a scale of 1-Novice to 4-Competent, for a total of 48 points. A score of 39 (80%) is considered competent.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Chaya, MD, Principal Investigator — University of Utah John A. Moran Eye Center
Locations (1):
- University of Utah John A. Moran Eye Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No